CLINICAL TRIAL: NCT05325593
Title: A Multicentre, Randomized, Open-label Study of Romiplostim Plus Dexamethasone vs Dexamethasone in Patients With Newly Diagnosed Primary Immune Thrombocytopenia
Brief Title: Romiplostim Plus Dexamethasone vs Dexamethasone in Patients With Newly Diagnosed Primary Immune Thrombocytopenia
Acronym: RODEX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RODEX; 2024-514147-28-00 (EU CTIS Number); 2021-006970-22 (EudraCT Number)
Record Dates: First submitted 2022-03-07; First posted 2022-04-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: Romiplostim; Dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- romiplostim plus dexamethasone (ROM + DEX) (Experimental): Dexamethasone 40 mg daily x 4 days only in the first cycle and subcutaneous romiplostim weekly for up to 12 months
  Romiplostim:
  1. The starting dose should be 3 mcg/kg/week. It could be start during de 4 days of dexamethasone.
  2. Patients will weekly receive dose increases of romiplostim in increments of 1 mcg/kg up to a maximum dose of 10 mcg/kg in an attempt to reach a target platelet count higher than 50x109/L.
  3. Otherwise, if platelets are lower than 50x109/L treatment with romiplostim will go on until Day 365 since randomization.
  Interventions: Drug: romiplostim plus dexamethasone
- Dexamethasone (DEX) (Active Comparator): Dexamethasone 40 mg daily x 4 days for up to 3 cycles every 14 to 28 days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: romiplostim plus dexamethasone — Patients will be reviewed weekly for 8 weeks (56 days). After Week 8, patients will be reviewed every 2 weeks (14 days) for 8 additional weeks and then monthly until Week 52 (365 days) from randomization.
  Other Names: ROM + DEX
  Arms: romiplostim plus dexamethasone (ROM + DEX)
Drug: Dexamethasone — Patients will be reviewed weekly until the completion of dexamethasone cycles and for a minimum of 8 weeks (56 days). After that, every 2 weeks (14 days) for 8 additional weeks and then monthly until Week 52 (365 days) from randomization.
  Other Names: DEX
  Arms: Dexamethasone (DEX)

SUMMARY:
Phase III, open-labeled, randomized and multicenter clinical trial to evaluate the superiority of romiplostim plus dexamethasone vs dexamethasone alone in patients with newly diagnosed primary immune thrombocytopenia

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the superiority of romiplostim plus dexamethasone versus dexamethasone alone in the treatment of primary immune thrombocytopenia, with sustained response to any ITP treatment and without World Health Organization grade 2 or higher bleeding, after six months from cessation of treatment.

Maximum time on treatment with romiplostim will be 12 months (365 days). Then, patients will be followed up for 6 additional months (180 days) after stopping romiplostim.

Clinical rules are included if romiplostim dose should be modified or finished. In case of dexamethasone, no dose adjustment is permitted.

The evaluation of romiplastim plus dexamethasone´s superiority in different periods and platelet count, proportion of patients with complete response (CR), global response (GR), early response (ER) and initial response (IR); time to loss of response (LoR), adverse events, quality of life and healthcare resources use are included as secondary objectives.

ELIGIBILITY:
Main inclusion criteria:

1. Age ≥ 18 years of age at the time of signing informed consent.
2. Newly diagnosis of primary ITP according to the International Working Group assessment [1] and previously untreated for ITP.
3. Platelet counts <30x109/L or ITP with platelet counts <50x109/L and concomitant bleeding symptoms.
4. Serum creatinine concentration ≤1.5 mg/dL.

Main exclusion criteria:

1. World Health Organization's performance status >2.
2. Previous therapy with rituximab (within 3 months previous of study enrollment), corticosteroids or, therapy with other immunomodulating agents within 1 month before of enrolment;,prior use of hematopoietic analogs and or fostamatinib for any other reason despite ITP three months before enrolment.
3. Previous use of romiplostim, polyethylene glycol-recombinant human megakaryocyte growth and development factor, Eltrombopag, recombinant human anti-thrombopoietin, or any platelet-producing agent three months before enrolment.
4. Alkylating agents within 8 weeks before the screening visit or anticipated use during the time of the proposed study.
5. Splenectomy within 3 months of the screening visit or planned splenectomy during study period.
6. Abnormal renal function (serum creatinine > 1.5 mg/dL).
7. Active hepatic disease (evidenced by alanine aminotransferase [ALT] or aspartate aminotransferase [AST] levels >5 times the upper limit of normal (it will only be necessary to determine one of the two transaminases
8. Severe chronic liver disease as evidenced by, but not limited to, any of the following: International Normalized Ratio >1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices.
9. Patients with known immunoglobulin M seropositive tests for cytomegalovirus and/or Epstein-Barr virus in the previous month.
10. Patients with an active viral infection at screening with: Hepatitis B Virus, Hepatitis C Virus, detectable virus charge of HIV.
11. Intolerance to dexamethasone.
12. History of a bone marrow stem cell disorder.
13. Active or prior malignancy except adequately treated (ie, complete surgical excision with negative margins) basal cell carcinoma.
14. History of helicobacter pylori by urea breath test or stool antigen test within 6 months of enrollment, if available.
15. History of myelodysplastic syndrome, systemic lupus erythematosus, or autoimmune cytopenia.
16. History of antiphospholipid antibody syndrome.
17. History of disseminated intravascular coagulation, hemolytic uremic syndrome, or thrombotic thrombocytopenic purpura.
18. History of deep or superficial venous thromboembolism in the last 12 months or stroke, acute ischaemic heart disease or acute peripheral vascular disease in the last 6 months.
19. Hypersensitivity to any recombinant Escherichia coli-derived product (eg, Infergen, Neupogen, Somatropin, and Actimmune) or known sensitivity to any of the products to be administered during dosing
20. Currently enrolled in another investigational device or drug study or < 30 days since ending another investigational device or drug studies, or receiving other investigational agents.
21. Will have any other investigational procedures performed while enrolled in this clinical study.
22. Pregnant or breastfeeding, or planning to become pregnant or breastfeed during treatment or within 1 month after the end of treatment.
23. Female subject of childbearing potential is not willing to use, in combination with her partner, an acceptable method of effective contraception during treatment and for 1 month after the end of treatment. Females of childbearing potential should only be included after a negative, pregnancy test.
24. Will not be available for protocol-required study visits, to the best of the subject's and investigator's knowledge.
25. Any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures.
26. Other serious comorbidities at investigator criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2026-10-24 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving sustain response out of treatment with platelets higher or equal than 30x109/L for 6 months (Sustained Response Off any ITP Treatment) | 180 days after treatment withdrawal
  Proportion of patients with platelets higher or equal than 50x109/L in the absence of any ITP treatment including any rescue treatment for at least 6 consecutive months (≥180 days) from treatment cessation and without World Health Organization grade 2 or more bleeding

SECONDARY OUTCOMES:
Proportion of patients achieving sustain response out of treatment with platelets higher or equal than 30x109/L for 6 months in the absence of any ITP treatment including any rescue treatment. | 180 days after treatment withdrawal
  Proportion of patients with platelets higher or equal than 30x109/L in the absence of any ITP treatment including any rescue treatment for at least 6 consecutive months (≥180 days) from treatment cessation and without World Health Organization grade 2 or more bleeding.
Proportion of patients achieving sustain response out of treatment with platelets higher or equal than 30x109/L for 12 months in the absence of any ITP treatment including any rescue treatment. | 365 days after treatment withdrawal
  Proportion of patients with platelets higher or equal than 30x109/L in the absence of any ITP treatment including any rescue treatment for at least 12 consecutive months (≥365 days) from treatment cessation and without World Health Organization grade 2 or more bleeding.
Proportion of patients achieving sustain response out of treatment with platelets higher or equal than 50x109/L for 12 months in the absence of any ITP treatment including any rescue treatment. | 365 days after treatment withdrawal
  Proportion of patients with platelets higher or equal than 50x109/L in the absence of any ITP treatment including any rescue treatment for at least 12 consecutive months (≥365 days) from treatment cessation and without World Health Organization grade 2 or more bleeding.
Proportion of patients with early response (ER) | Day 7
  Proportion of patients with platelet count higher or equal than 30x109/L and at least double than baseline.
Proportion of patients with initial response (IR) | Day 30
  Proportion of patients with platelet count higher or equal than 30x109/L
Proportion of patients with complete response (CR) | Day 180, Day 365, Day 545
  Patients with platelet count ≥100x109/L and absence of bleeding symptoms.
Proportion of patients with response (R) | Day 180, Day 365, Day 545
  Patients with platelet count between 100x109/L and 30x109/L and at least doubled from baseline and absence of bleeding symptoms.
Proportion of patients with global response (GR) | Day 180, Day 365, Day 545
  Patients with platelet count ≥100x109/L and absence of bleeding symptoms or platelet count between 100x109/L and 30x109/L and at least doubled from baseline and absence of bleeding symptoms.
Proportion of patients with targeted range (TR) | Day 180, Day 365, Day 545
  Patients with platelet count between ≥30x109/L and ≤400x109/L.
Time to loss of response (LoR) in patients who achieved response in both arms. | In every study visit, assessed up to 545 days
  Number of days from the first time the patient achieved a platelet count ≥30x109/L until platelet count dropped below 30x109/L measured on 2 occasions with more than 1 day apart or presence of bleeding
Proportion of patients requiring any rescue treatment | In every study visit, assessed up to 545 days
  Proportion of patients who need rescue treatments in each arm and total patients
Proportion and time to treatment failures | In every study visit, assessed up to 545 days
  Proportion of patients who need rescue treatments and And the number of days they needed treatment
Proportion of patients with adverse events (AEs), including serious adverse events (SAEs) and laboratory safety parameters. | In every study visit, assessed up to 545 days
  AEs will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Bleeding events will be carefully monitored
Changes in patients bleeding | Screning, Day 1, Week 8, Week 12, Moth 6, Moth 12 and End of study Visit
  For the assessment of the of the patients' bleeding will be used immune thrombocytopenia-bleeding assessment tool (ITP-BAT): bleeding signs/symptoms are grouped in three domains (skin, visible mucosae and organs) and is graded from 0 (No) to 4.
Changes in patients' quality of life- Short Form-36 Health Survey | Day 1, Week 8, Day 180, Day 365 and Day 545
  For the assessment of the quality of life during the study will be used Short-Form-36 Health Survey: is a 36-item scale constructed to survey health-related 8 domains: limitations in physical activities due to health problems; limitations in social activities due to physical or emotional problems; limitations unusual role activities due to physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations unusual role activities due to emotional problems; vitality (energy and fatigue); and general health perceptions.
Changes in patients' quality of life- FACIT-F | Day 1, Week 8, Day 180, Day 365 and Day 545
  For the assessment of the quality of life during the study will be used FACIT-F (Fatigue Scale): is a short scale, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week.The level of fatigue is measured by recording item responses ona 4-point Likert scale ranging from 0 "not at all" to 4 "very much.
Changes in patients' quality of life- ITP-Patient Assessment Questionnaire | Day 1, Week 8, Day 180, Day 365 and Day 545
  For the assessment of the quality of life during the study will be used ITP-Patient Assessment Questionnaire): is a disease-specific instrument that was designed to measure the QoL of adult patients with immune thrombocytopenia. The instrument comprises 38 items completed by male respondents and 44 items completed by female respondents.
Healthcare resources use (HRU) | In every study visit, assessed up to 545 days
  The data collected may be used to conduct exploratory economic analyses and may include:
  * Number of outpatient visits,
  * Number of home health care
  * Number of Hospitalization
  * Duration of medical care visits (days)
  * Number of Emergency room visits
  * Number of diagnostic procedures
  * Number of medical care visits
Loss of productivity | In every study visit, assessed up to 545 days
  Number of days of absenteeism from school or work and associated cost
Maximum number of consecutive days with platelet response | In every study visit, assessed up to 545 days
  - The maximum number of consecutive days with platelet count between 100x109/L and 30x109/L in the total sample and in the absence of any rescue treatment
Maximum number of consecutive days with platelet complete response (CR) | In every study visit, assessed up to 545 days
  - The maximum number of consecutive days with platelet count ≥100x109/L in the total sample and in the absence of any rescue treatment
Maximum number of consecutive days with platelet global response (GR) | In every study visit, assessed up to 545 days
  The maximum number of consecutive days with platelet count ≥100x109/L or platelet count between 100x109/L and 30x109/L in the total sample and in the absence of any rescue treatment
Maximum number of consecutive days with platelet targeted range (TR) | In every study visit, assessed up to 545 days
  The maximum number of consecutive days with platelet count between ≥30x109/L and ≤400x109/ L in the total sample and in the absence of any rescue treatment
Total number of days with platelet response | In every study visit, assessed up to 545 days
  The total number od days with platelet count ≥100x109/L in the total sample and in the absence of any rescue treatment
Total number of days with platelet complete response (CR) | In every study visit, assessed up to 545 days
  The total number od days with platelet count ≥100x109/L in the total sample and in the absence of any rescue treatment
Total number of days with platelet global response (GR | In every study visit, assessed up to 545 days
  The total number od days with platelet count ≥100x109/L or platelet count between 100x109/L and 30x109/L in the total sample and in the absence of any rescue treatment
Total number of days with platelet targeted range (TR) | In every study visit, assessed up to 545 days
  The total number od days with platelet count between ≥30x109/L and ≤400x109/ L in the total sample and in the absence of any rescue treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Bradbury, Principal Investigator — Centre for Trials Research College of Biomedical & Life Sciences Cardiff University
Locations (30):
- Italy (6):
  - IRCCS AOU di Bologna, Seràgnoli Institute of Hematology, Bologna
  - ASST Fatebenefratelli Sacco - Ospedale L. Sacco, Milan
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I / SAPIENZA Universitá di Roma, Rome
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Spain (15):
  - Hospital del Mar, Barcelona, Barcelona
  - Centre Sociosanitari Sant Jordi de la Vall D'Hebron, Barcelona, Barcelona
  - Complejo Asistencial Universitario de Burgos, Burgos, Burgos
  - Complejo Hospitalario Universitario A Coruña, A Coruña, Coruña
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Compejo Hospitalario La Paz, Madrid, Madrid
  - Hospital Universitario Fundación Alcorcon, Madrid, Madrid
  - Hospital Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Complejo Asistencial Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitario y Pilitécnico La Fe, Valencia, Valencia
  - Complejo Asistencial Son Espases, Palma de Mallorca
- United Kingdom (9):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol and Weston NHS Trust, Bristol
  - Haemophilia and Thrombosis Centre, Kent & Canterbury Hospital, Kent & Canterbury Hospital, Ethelbert Road, Canterbury, CT1 3NG, England, UK, Canterbury
  - Greater Glasgow and Clyde Health Board, London
  - Haematology, Royal Victoria Infirmary, Newcastle
  - Norfolk & Norwich University Hospital Trust, Norwich
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - "Haematology, Derriford Hospital, University Hospitals Plymouth NHS Trust, Plymouth
  - Torbay and South Devon NHS Foundation Trust, Torquay

IPD SHARING:
Plan to Share IPD: Yes
The results will be shared with the investigators involved in the study, and will be shared when the analysis of the results is performed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Along the study
Access Criteria: Direct collaborators within the study